CLINICAL TRIAL: NCT03574311
Title: A Phase IV Double-blind, Randomised, Parallel Group Comparison of the Efficacy and Safety of Preoperative Intravenous Ferric Carboxymaltose and Placebo in the Treatment of Patients Undergoing Elective or Urgent Cardiac Surgery
Brief Title: Preoperative Intravenous Ferric Carboxymaltose and Placebo in the Treatment of Patients Undergoing Cardiac Surgery
Acronym: PREFER-CABG
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Turku University Hospital (Other Government)
Collaborators: Vifor Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PREFER-CPB01
Record Dates: First submitted 2018-06-14; First posted 2018-06-29 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Coronary Artery Disease; Postoperative Complications; Aortic Valve Stenosis; Mitral Valve Disease; Aortic Aneurysm, Thoracic
Keywords: CABG; cardiac surgery; blood transfusion; intravenous iron; postoperative infection
MeSH Terms: conditions — Coronary Artery Disease; Postoperative Complications; Aortic Valve Stenosis; Aortic Aneurysm, Thoracic | interventions — ferric carboxymaltose

STUDY DESIGN:
Intervention Model Description: Randomized controlled 1:1
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double blinding, study drug administration by separate staff blinded from participant and investigators
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ferric carboxymaltose (Experimental): Preoperative 1000 mg intravenous single dose as 30 minute infusion
  Interventions: Drug: Ferric carboxymaltose
- Placebo (Placebo Comparator): Preoperative 100 ml saline as 30 minute infusion
  Interventions: Other: Physiological saline

INTERVENTIONS:
Drug: Ferric carboxymaltose — A single dose of drug or placebo is administered preoperatively to participants
  Arms: Ferric carboxymaltose
Other: Physiological saline — Single infusion 100 ml physiological saline infusion preoperatively
  Arms: Placebo

SUMMARY:
This study evaluates the efficacy and safety of single dose preoperative ferric carboxymaltose in the prevention of postoperative infections and blood transfusions in patients scheduled for cardiac surgery. Half of the patients will receive ferric carboxymaltose and half of the patients physiological saline solution as placebo.

ELIGIBILITY:
Inclusion criteria:

1. Patients presenting with cardiac disease requiring surgical operation
2. Open heart surgery is considered the best appropriate treatment strategy according to the current guidelines.

   * significant three vessel disease
   * left main disease ± single, two or three vessel disease
   * two-vessel disease with proximal LAD stenosis
   * coronary artery disease requiring revascularization not amenable to percutaneous coronary intervention
   * Aortic valve disease requiring aortic valve surgery
   * Mitral valve disease requiring surgical mitral surgery
   * Combined surgery for revascularization and valve disease
   * surgery of ascending aorta
3. Have provided signed written informed consent

Exclusion Criteria:

1. Age < 35 years
2. Patients requiring , emergency or salvage cardiac surgical operation
3. Participation in another clinical study or treatment with another investigational product 30 days prior to randomization
4. Moribund patient not expected to survive surgery 12 months after surgery
5. Active malignant disease with a short life expectancy, not eligible for surgery
6. Hemoglobin levels > 155 g/dL for women and >167 g/dl for men (upper reference limits for TYKSlab)
7. Ferritin levels >150 ug/l for women and >400 ug/l for men.
8. Renal dialysis therapy for chronic renal failure or severe preoperative renal impairment (eGFR<30ml/min).
9. Study treatment can't be infused during the required time window: minimum 48 hours and maximum 21 days before the operation.
10. Ongoing oral or parenteral iron medication at the time of randomization
11. Iron or haemoglobin metabolism or synthesis disorders
12. Primary or secondary hemochromatosis (in males and postmenopausal females, a serum ferritin value of over 300 ng/mL (670 pmol/L); and in premenopausal females, a serum ferritin value of over 150[17] or 200[18] ng/mL (330 or 440 pmol/L) indicates iron overload).
13. Porphyria cutanea tarda.
14. Liver failure (Child-Pugh class B or C).
15. Pregnancy.
16. Body weight less than 50kg.
17. Ongoing antibiotic treatment other than prophylactic urine tract infection antibiotics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2018-10-02 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of allogeneic blood transfusion and/or nosocomial infection | 0-90 days
  Composite of transfused red blood cell units and/or nosocomial infection

SECONDARY OUTCOMES:
Mortality | 0-90 days
  All-cause mortality
ICU/CCU days | 0-90 days
  Days in the ICU (intensive care unit) and/or CCU (cardiac care unit)
Perioperative myocardial infarction | 3 days
  MI (myocardial infarction) assessed by postoperative CK-Mbm or Troponin t levels
Length of stay | 0-90 days
  Days in hospital
Days on vasoactive drugs | 0-90 days
  Days on vasopressors (e.g. epinephrine, norepinephrine, milrinone etc.)
Ventilator free days | 0-90 days
  Days not on ventilator (intubated or non-invasive ventilation)
AKI (acute kidney injury) | 0-90 days
  Rate of acute renal failure
New onset atrial fibrillation (AF) or flutter | 0-90 days
  New AF or flutter (i.e. patient without previous history of AF/flutter) assessed from ECG-telemetry during index hospitalization or ECG-verified AF/flutter after discharge
Acute heart failure | 90 days
  Acute congestive heart failure (diagnosed by a clinician) requiring hospitalization
Worsening heart failure | 0-90 days
  Worsening to NYHA -class (New York Heart Association) III/IV or readmission for heart failure
Health related quality of life | 12 months
  Assessed with self-reporting questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Turku University Hospital, Turku, Finland

IPD SHARING:
Plan to Share IPD: No